CLINICAL TRIAL: NCT01240863
Title: A 12-Week, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Hydrocodone Bitartrate Extended-Release Tablets (CEP-33237) at 15 to 90 mg Every 12 Hours for Relief of Moderate to Severe Pain in Patients With Osteoarthritis or Low Back Pain Who Require Opioid Treatment for an Extended Period of Time
Brief Title: Study to Evaluate the Efficacy and Safety of Hydrocodone Bitartrate Extended-Release Tablets (CEP-33237) for Relief of Moderate to Severe Pain in Patients With Osteoarthritis or Low Back Pain Who Require Opioid Treatment for an Extended Period of Time
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C33237/3079
Record Dates: First submitted 2010-11-10; First posted 2010-11-15 (Estimated); Results first posted 2017-06-05 (Actual); Last update posted 2017-06-05 (Actual); Status verified 2017-06

CONDITIONS: Chronic Pain
Keywords: osteoarthritis; low back pain; Moderate to Severe Pain
MeSH Terms: conditions — Chronic Pain; Osteoarthritis; Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Participants were administered hydrocodone ER tablets at dosages of 15, 30, 45, 60, or 90 mg every 12 hours at the dosage deemed successful for managing their pain during the titration period. During the treatment period, participants were administered placebo tablets every 12 hours that matched the dosage deemed successful for managing their pain during the titration period. A step-wise, double-blind schedule to tamper off active drug was implemented during the first 2 weeks of the 12-week, double-blind, placebo-controlled treatment period to reduce the risk of withdrawal effects in participants randomly assigned to placebo.
  Interventions: Drug: Hydrocodone ER; Drug: Placebo
- Hydrocodone ER (Experimental): Participants were administered hydrocodone ER tablets at dosages of 15, 30, 45, 60, or 90 mg every 12 hours at the dosage deemed successful for managing their pain during the titration period. During the 12-week, double-blind, placebo-controlled treatment period, participants randomly assigned to hydrocodone ER were administered tablets every 12 hours at the dosage deemed successful for managing their pain during the titration period.
  Interventions: Drug: Hydrocodone ER

INTERVENTIONS:
Drug: Hydrocodone ER — During the open-label, titration period, all participants were administered hydrocodone ER tablets at dosages of 15, 30, 45, 60, or 90 mg every 12 hours to identify a dosage deemed successful for managing their pain.
  Hydrocodone ER was taken by participants randomized to the hydrocodone ER treatment arm during the double-blind treatment period at the dose level identified during the titration period.
  Participants were instructed to take tablets with a glass of water on an empty stomach at least 1 hour before or 2 hours after eating.
  Other Names: CEP-33237; Hydrocodone bitartrate extended-release
Drug: Placebo — Placebo matching the active drug dose identified during the titration period was taken by participants randomized to the placebo treatment arm during the double-blind treatment period.
  Participants were instructed to take intervention with a glass of water on an empty stomach at least 1 hour before or 2 hours after eating.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate efficacy of hydrocodone extended-release (ER) tablets compared with placebo in alleviating moderate to severe pain in patients with osteoarthritis or low back pain as assessed by the weekly Average Pain Intensity (API) at week 12.

DETAILED DESCRIPTION:
The study consisted of a screening period of approximately 7 to 14 days, an open label titration period of up to 6 weeks, and a double blind treatment period of 12 weeks.

Participants entered the open label titration period and received hydrocodone ER tablets beginning with 15 mg every 12 hours for 3 to 7 days. The objective of the open label titration period was to find the successful dose of hydrocodone ER tablets that produced stable pain relief (defined as an Average Pain Intensity (API) score of 4 or less on the 11-point numerical rating scale for either 3 consecutive days or 3 out of 5 consecutive days while the patient was maintained on the same dose of study drug for up to 7 days). Patients returned to the study center prior to each dose adjustment.

Participants who met the criterion of a stabilized dose were randomly assigned into the 12 week, double blind, placebo controlled treatment period on the final day of the open label titration period (baseline visit). Patients began treatment with double blind study drug at the effective dose of hydrocodone ER tablets achieved during the titration period or matching placebo. Rescue medication was permitted in addition to the study drug during the double blind treatment period.

ELIGIBILITY:
Inclusion Criteria:

* The patient is able to speak English and is willing to provide written informed consent, including a written opioid agreement, to participate in this study.
* The patient must be willing and able to successfully self-administer the study drug, comply with study restrictions, complete the electronic diary, and return to the clinic for scheduled study visits as specified in this protocol.
* Women of childbearing potential (not surgically sterile or 2 years postmenopausal), must use a medically accepted method of contraception and must agree to continue use of this method for the duration of the study and for 30 days after participation in the study, and have a negative pregnancy test at screening.
* The patient has pain of at least 3 months' duration associated with osteoarthritis or low back pain.
* The patient reports an average pain intensity score, over the prior 24 hours, of 5 or more on the 11-point numerical rating scale.
* If the patient is receiving physical therapy, biofeedback therapy, acupuncture therapy, or herbal remedies, these therapies must remain unchanged during the study.
* The patient must not participate in other study involving an investigational agent while enrolled into the present study.

Exclusion Criteria:

* The patient has known or suspected hypersensitivities, allergies, or other contraindications to any ingredient in the study drug.
* The patient has a recent history (within 5 years) or current evidence of alcohol or other substance abuse with the exception of nicotine or caffeine.
* The patient has medical or psychiatric disease that, in the opinion of the investigator, would compromise collected data.
* The patient is taking a total (ie, around-the-clock plus rescue medication) of more than 135 mg/day of oxycodone, or equivalent, during the 14 days prior to screening.
* The patient has a history of suicidality.
* The patient is expected to have surgery during the study.
* The patient's primary painful condition under study is related to any source of chronic pain other than osteoarthritis or low back pain.
* The patient is pregnant or lactating.
* The patient has active malignancy.
* The patient has human immunodeficiency virus (HIV).
* In the judgment of the investigator, the patient has any clinically significant deviation from normal in the physical examination and/or clinical laboratory test values.
* The patient has cardiopulmonary disease that would, in the opinion of the investigator, significantly increase the risk of treatment with opioids.
* The patient has participated in a study involving an investigational drug in the previous 30 days.
* The patient has received a monoamine oxidase inhibitor (MAOI) within 14 days before the first treatment with study drug.
* The patient has any other medical condition or is receiving concomitant medication/therapy (e.g., regional nerve block) that would, in the opinion of the investigator, compromise the patient's safety or compliance with the study protocol, or compromise collected data.
* The patient is involved in active litigation in regard to the pain currently being treated.
* The patient has a positive urine drug screen (UDS) that is not medically explainable.
* The investigator feels that the patient is not suitable for the study for any reason.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 391 (Actual)
Dates: Start 2010-11; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sponsor's Medical Expert, MD, Study Director — Cephalon
Locations (72):
- United States (72):
  - Horizon Research Group LLC, Mobile, Alabama
  - Radiant Research, Inc., Chandler, Arizona
  - Radiant Research, Inc., Scottsdale, Arizona
  - Radiant Research Inc., Tucson, Arizona
  - Physician Alliance Research Center, Anaheim, California
  - Associated Pharmaceutical Research Center, Inc., Buena Park, California
  - Providence Clinical Research, Burbank, California
  - Synergy Clinical Research, Escondido, California
  - Research Center of Fresno, Inc., Fresno, California
  - Pacific Coast Pain Management Center, Laguna Hills, California
  - South Orange County Surgical Medical Group, Laguna Hills, California
  - Robert M. Karns, MD A Medical Corporation, Los Angeles, California
  - Accelovance, Inc., San Diego, California
  - Radiant Research, Inc., Santa Rosa, California
  - Bayview Research Group, LLC, Valley Village, California
  - Radiant Research, Inc, Denver, Colorado
  - Clinical Research of West Florida, Inc., Clearwater, Florida
  - Avail Clinical Research, LLC, DeLand, Florida
  - International Research Associates, LLC, Miami, Florida
  - Compass Research, Orlando, Florida
  - Radiant Research, Inc., Pinellas Park, Florida
  - Gold Coast Research LLC, Plantation, Florida
  - Sarasota Pain Medicine Research LLC, Sarasota, Florida
  - Clinical Research of West Florida, Inc., Tampa, Florida
  - Drug Studies America, Marietta, Georgia
  - Georgia Institute for Clinical Research, LLC, Marietta, Georgia
  - Better Health Clinical Research, Inc., Newnan, Georgia
  - Millennium Pain Center, Bloomington, Illinois
  - Medex Healthcare Research, Inc., Chicago, Illinois
  - Rehabilitation Associates of Indiana, Indianapolis, Indiana
  - International Clinical Research, Inc., Leawood, Kansas
  - Community Research, Crestview, Kentucky
  - The Pain Treatment Center of the Bluegrass, Lexington, Kentucky
  - Horizon Research Group, LLC, Baton Rouge, Louisiana
  - WK River Cities Clinical Research Center, Shreveport, Louisiana
  - MidAtlantic Pain Medicine Center, Pikesville, Maryland
  - Beacon Clinical Research, LLC, Brockton, Massachusetts
  - HealthCare Research, Florissant, Missouri
  - Medex Healthcare Research Inc., St Louis, Missouri
  - Sundance Clinical Research, LLC, St Louis, Missouri
  - Meridian Clinical Research, Omaha, Nebraska
  - Clinical Research Center of Nevada, Las Vegas, Nevada
  - Advanced Pain Consultants, Voorhees Township, New Jersey
  - Upstate Clinical Research Associates, Williamsville, New York
  - Wake Research Associates, Raleigh, North Carolina
  - Radiant Research, Inc, Akron, Ohio
  - Sterling Research Group, Ltd., Cincinnati, Ohio
  - Community Research, Inc, Cincinnati, Ohio
  - Rapid Medical Research, Cleveland, Ohio
  - Columbus Clinical Research, Columbus, Ohio
  - SP Research, Oklahoma City, Oklahoma
  - Pain Research of Oregon, Eugene, Oregon
  - Summit Research Network Inc., Portland, Oregon
  - Brandywine Clinical Research, Downingtown, Pennsylvania
  - Tipton Medical and Diagnostic Center, Tipton, Pennsylvania
  - AMH Feasterville Family Health Care Center, Trevose, Pennsylvania
  - Clinical Research Center of Reading, Wyomissing, Pennsylvania
  - Omega Medical Research, Warwick, Rhode Island
  - Radiant Research Inc., Anderson, South Carolina
  - Greenville Pharmaceutical Research, Greenville, South Carolina
  - Radiant Research, Inc, Greer, South Carolina
  - Trident Institute of Medical Research, LLC, North Charleston, South Carolina
  - South Carolina Pharmaceutical Research, Spartanburg, South Carolina
  - KRK Medical Research, Dallas, Texas
  - Radiant Research Dallas, Dallas, Texas
  - Renaissance Clinical Research & Hypertension of Texas, PLLC, Dallas, Texas
  - Medstar Clinical Research, Houston, Texas
  - Benchmark Research, San Angelo, Texas
  - DCT-Sugarland, LLC, Sugar Land, Texas
  - Hillcrest Family Health Centers, Waco, Texas
  - Aspen Clinical Research, LLC, Orem, Utah
  - Lifetree Clinical Research, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 519 patients with osteoarthritis or low back pain were screened for enrollment into the study; of these, 391 patients at 71 centers in the US met entry criteria and were enrolled into the titration period of the study.
Pre-assignment Details: Of the 389 patients enrolled and treated during the titration period, 294 (75%) patients identified a successful dose and therefore completed the open-label titration period, and were randomly assigned to receive hydrocodone extended-release (ER) tablets (146 patients) or placebo (148 patients) in the double-blind treatment period.
Groups:
- Hydrocodone ER (Open-Label Titration Period): All enrolled participants entered the open label titration period and received hydrocodone extended release (ER) tablets beginning with 15 mg every 12 hours for 3 to 7 days. Dosages were titrated upward until pain was effectively controlled. If an effective dosage between 15 mg - 90 mg twice a day was not identified within 6 week, the participant was withdrawn.
- Placebo (Double-blind Treatment Period): Participants were administered placebo tablets twice a day that matched the dosage deemed successful for managing their pain during the titration period. A step wise, double-blind tapering schedule was implemented during the first 2 weeks of the 12 week, double blind, placebo controlled treatment period to reduce the risk of withdrawal effects in patients randomly assigned to placebo.
- Hydrocodone ER (Double-blind Treatment Period): Participants were administered hydrocodone ER tablets at a dosage deemed successful for managing their pain during the titration period. Dosages of 15, 30, 45, 60, or 90 mg every 12 hours were given for 12 weeks during the double-blind period.
Period: Open-label Titration Period
Arm/Group | Hydrocodone ER (Open-Label Titration Period) | Placebo (Double-blind Treatment Period) | Hydrocodone ER (Double-blind Treatment Period)
Started | 391 | 0 | 0
Safety Analysis Set | 389 | 0 | 0
Completed | 294 | 0 | 0
Not Completed | 97 | 0 | 0
Not completed — Adverse Event | 47 | 0 | 0
Not completed — Lack of Efficacy | 19 | 0 | 0
Not completed — Withdrawal by Subject | 9 | 0 | 0
Not completed — Protocol Violation | 7 | 0 | 0
Not completed — Noncompliance to study drug admin | 3 | 0 | 0
Not completed — Noncompliance to study procedures | 3 | 0 | 0
Not completed — Dropped out prior to dosing | 2 | 0 | 0
Not completed — Other | 7 | 0 | 0
Period: Double-blind Treatment Period (12 Weeks)
Arm/Group | Hydrocodone ER (Open-Label Titration Period) | Placebo (Double-blind Treatment Period) | Hydrocodone ER (Double-blind Treatment Period)
Started | 0 | 148 | 146
Full Analysis and Safety Analysis Sets | 0 | 147 | 146
Completed | 0 | 102 | 94
Not Completed | 0 | 46 | 52
Not completed — Adverse Event | 0 | 4 | 10
Not completed — Lack of Efficacy | 0 | 17 | 5
Not completed — Withdrawal by Subject | 0 | 3 | 5
Not completed — Protocol Violation | 0 | 9 | 14
Not completed — Noncompliance to study drug admin | 0 | 9 | 11
Not completed — Noncompliance to study procedures | 0 | 2 | 2
Not completed — Other | 0 | 1 | 5
Not completed — Physician Decision | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Randomized participants
Groups:
- Placebo (Double-blind Treatment Period): Participants were administered placebo tablets every 12 hours that matched the dosage deemed successful for managing their pain during the titration period. A step wise, double-blind tapering schedule was implemented during the first 2 weeks of the 12 week, double blind, placebo controlled treatment period to reduce the risk of withdrawal effects in patients randomly assigned to placebo.
- Total: Total of all reporting groups
Arm/Group | Placebo (Double-blind Treatment Period) | Hydrocodone ER (Double-blind Treatment Period) | Total
Number analyzed (Participants) | 148 | 146 | 294
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.7 (12.09) | 53.6 (10.38) | 53.1 (11.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 87 | 175
  Male | 60 | 59 | 119
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 105 | 115 | 220
  Black | 41 | 28 | 69
  Other | 2 | 3 | 5
  Asian | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 9 | 12
  Non-Hispanic and non-Latino | 144 | 137 | 281
  Unknown | 1 | 0 | 1
Age group [Count of Participants; unit: Participants]
  <=65 years | 133 | 126 | 259
  >65 years | 15 | 20 | 35
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 32.8 (7.33) | 33.0 (8.16) | 32.9 (7.74)
Type of Pain [Count of Participants; unit: Participants]
  Low back pain | 107 | 104 | 211
  Osteoarthritis | 41 | 42 | 83
Duration since Diagnosis [Mean (Standard Deviation); unit: years] | 12.5 (9.06) | 12.1 (9.97) | 12.3 (9.51)
Participants on Opioid Therapy [Count of Participants; unit: Participants]
  On opioid therapy | 103 | 100 | 203
  Not on opioid therapy | 45 | 46 | 91
Duration of Opioid Therapy [Mean (Standard Deviation); unit: years] — Population: Includes participants with duration of opioid therapy data available.
  years
    number analyzed (Participants) | 103 | 100 | 203
    (all) | 4.1 (4.90) | 3.9 (4.76) | 4.0 (4.82)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 12 in Weekly Average Pain Intensity (wAPI)
Description: The primary efficacy variable was the change from baseline to week 12 in the wAPI. The API over the previous 24 hours, based on the 11-point Numerical Rating Scale (NRS 11), was collected daily by e-diary. The Week 12 wAPI scores from the previous 7 days were calculated for each study visit and averaged. The baseline wAPI score was calculated by averaging API scores from 3 to 12 days when the successful dose of hydrocodone extended release was confirmed at the end of the open label titration period, before patients were randomly assigned study drug. In the case of missing week-12 data due to early withdrawal from the study, or excessive rescue medication usage, the wAPI for week 12 was imputed.
  The Numeric Rating Scale (NRS-11) is an 11-point scale for patient self-reporting of pain on a Likert-type scale in which 0 is no pain and 10 is the worst pain imaginable. Negative change from baseline values indicate lessening in pain intensity.
Time Frame: Baseline (end of Open-Label Titration Period), Week 12 of Double-blind Treatment Period
Population: Full analysis set (FAS). One placebo patient was withdrawn from the study prior to receiving drug in the Double-blind Treatment period and is not included in the FAS. In the case of missing week-12 data due to early withdrawal from the study, or excessive rescue medication usage, the wAPI for week 12 was imputed.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo (Double-blind Treatment Period) | Hydrocodone ER (Double-blind Treatment Period)
Number analyzed (Participants) | 147 | 146
units on a scale | 0.14 (0.169) | -0.22 (0.176)
Statistical Analysis 1: Comparison: Placebo (Double-blind Treatment Period) vs Hydrocodone ER (Double-blind Treatment Period); Test type: Superiority or Other; p = 0.134, ANCOVA — statistical significance level of 0.05; Treatment and stratification (opioid naïve/opioid experienced) factors as the fixed effects; screening and baseline APIs as covariates; Mean Difference (Final Values) = 0.35, 95% CI 2-sided [-0.11 to 0.82] — placebo - hydrocodone

2. Secondary Outcome: Percentage of Participants Withdrawn From the Study During the Double-Blind Treatment Period By Reason
Description: Percentage of participants who withdrew from the study during the double-blind treatment period. Withdrawal is due to any cause, including lack of efficacy.
Time Frame: Day 1 to Week 12 of the double-blind treatment period
Population: Full analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Double-blind Treatment Period) | Hydrocodone ER (Double-blind Treatment Period)
Number analyzed (Participants) | 147 | 146
percentage of participants
  Total withdrawn from study period | 31 | 36
  Lack of efficacy | 12 | 3
  Adverse event | 3 | 7
  Consent withdrawn | 2 | 3
  Lost to follow-up | 0 | 0
  Protocol violation | 6 | 10
  Noncompliance to study procedures | 1 | 1
  Noncompliance to study drug admin | 6 | 8
  Other | 1 | 3

3. Secondary Outcome: Kaplan-Meier Estimates for Time to Discontinuation From the Study
Description: Kaplan-Meier estimates for time to discontinuation from the study (due to any cause) was calculated as the number of days since participants were randomly assigned to study drug treatment, ie, the difference between the date the participants withdrew and the date participants were randomly assigned to study drug treatment. The censoring flag was set to 0 if a participant was withdrawn from study drug treatment early and was set to 1 if the participant completed the 12 week treatment period. Censoring time was calculated as the difference of treatment completion date (ie, date of last study drug administration) and date participant was randomly assigned to study drug treatment.
Time Frame: Day 1 to Week 12 of the double-blind treatment period
Population: Full analysis set
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Placebo (Double-blind Treatment Period) | Hydrocodone ER (Double-blind Treatment Period)
Number analyzed (Participants) | 147 | 146
days | 99 [48 to 99] | NA [35 to NA] — not estimable due to low rate of discontinuation

4. Secondary Outcome: Participants With a Weekly Average Pain Intensity (wAPI) Increase From Baseline Exceeding 33%
Description: The API over the previous 24 hours, based on the 11-point Numerical Rating Scale (NRS 11), was collected daily by e-diary. The wAPI scores from the previous 7 days were calculated for each study visit and averaged. The baseline wAPI score was calculated by averaging API scores from 3 to 12 days when the successful dose of hydrocodone extended release was confirmed at the end of the open label titration period, before patients were randomly assigned study drug.
  The Numeric Rating Scale (NRS-11) is an 11-point scale for patient self-reporting of pain on a Likert-type scale in which 0 is no pain and 10 is the worst pain imaginable.
Time Frame: Baseline (end of Open-Label Titration Period), Weeks 1, 2, 4, 8, and 12 of the Double-blind treatment period
Population: Full analysis set. Participants contributing to each time point are included in the number analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Double-blind Treatment Period) | Hydrocodone ER (Double-blind Treatment Period)
Number analyzed (Participants) | 147 | 146
Participants
  Week 1 | 14 | 13
  Week 2: number analyzed (Participants) | 140 | 134
  Week 2 | 31 | 15
  Week 4: number analyzed (Participants) | 128 | 126
  Week 4 | 32 | 17
  Week 8: number analyzed (Participants) | 111 | 106
  Week 8 | 26 | 9
  Week 12: number analyzed (Participants) | 98 | 96
  Week 12 | 24 | 11

5. Secondary Outcome: Participants With a Weekly Average Pain Intensity (wAPI) Increase From Baseline Exceeding 50%
Description: as for outcome 4
Time Frame: Baseline (end of Open-Label Titration Period), Weeks 1, 2, 4, 8, and 12 of the Double-blind treatment period
Population: Full analysis set. Participants contributing to each time point are included in the number analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Double-blind Treatment Period) | Hydrocodone ER (Double-blind Treatment Period)
Number analyzed (Participants) | 147 | 146
Participants
  Week 1 | 7 | 9
  Week 2: number analyzed (Participants) | 140 | 134
  Week 2 | 16 | 9
  Week 4: number analyzed (Participants) | 128 | 126
  Week 4 | 19 | 9
  Week 8: number analyzed (Participants) | 111 | 106
  Week 8 | 20 | 6
  Week 12: number analyzed (Participants) | 98 | 96
  Week 12 | 15 | 6

6. Secondary Outcome: Weekly Average Pain Intensity (wAPI) Scores During the Double-blind Treatment Period
Description: as for outcome 4
Time Frame: Baseline (end of Open-Label Titration Period), Weeks 1, 2, 4, 8, and 12 of the Double-blind treatment period
Population: Full analysis set. Participants contributing to each time point are included in the number analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo (Double-blind Treatment Period) | Hydrocodone ER (Double-blind Treatment Period)
Number analyzed (Participants) | 147 | 146
units on a scale
  Baseline | 3.75 (0.903) | 3.79 (0.981)
  Week 1 | 3.73 (1.319) | 3.67 (1.291)
  Week 2: number analyzed (Participants) | 140 | 134
  Week 2 | 3.89 (1.498) | 3.58 (1.433)
  Week 4: number analyzed (Participants) | 128 | 126
  Week 4 | 3.78 (1.702) | 3.48 (1.447)
  Week 8: number analyzed (Participants) | 111 | 106
  Week 8 | 3.68 (1.823) | 3.16 (1.461)
  Week 12: number analyzed (Participants) | 98 | 96
  Week 12 | 3.61 (1.783) | 3.30 (1.638)

7. Secondary Outcome: Weekly Average Worst Pain Intensity (WPI) Scores During the Double-blind Treatment Period
Description: The WPI was recorded by the patient in the e-diary daily throughout the study, based on the Numeric Rating Scale (NRS-11). Participants were asked to select the number that best described their WPI over the previous 24 hours. Values were averaged for each week.
  The Numeric Rating Scale (NRS-11) is an 11-point scale for patient self-reporting of pain on a Likert-type scale in which 0 is no pain and 10 is the worst pain imaginable.
Time Frame: Baseline (end of Open-Label Titration Period), Weeks 1, 2, 4, 8, and 12 of the Double-blind treatment period
Population: Full analysis set. Participants contributing to each time point are included in the number analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo (Double-blind Treatment Period) | Hydrocodone ER (Double-blind Treatment Period)
Number analyzed (Participants) | 147 | 146
units on a scale
  Baseline | 4.75 (1.369) | 4.85 (1.265)
  Week 1 | 4.79 (1.776) | 4.79 (1.636)
  Week 2: number analyzed (Participants) | 140 | 134
  Week 2 | 5.02 (1.951) | 4.65 (1.781)
  Week 4: number analyzed (Participants) | 128 | 126
  Week 4 | 4.77 (2.099) | 4.55 (1.832)
  Week 8: number analyzed (Participants) | 111 | 106
  Week 8 | 4.57 (2.228) | 4.18 (1.892)
  Week 12: number analyzed (Participants) | 98 | 96
  Week 12 | 4.57 (2.210) | 4.22 (1.873)

8. Secondary Outcome: Clinician Assessment of Patient Function (CAPF) at Week 4
Description: Clinicians assessed participants across 5 dimensions:
  * Patients general activities
  * Patients walking ability
  * Patients ability to work/perform activities of daily living
  * Patients relationships with others
  * Patients enjoyment of life
  Assessments are rated on a 7-point scale, in which 1 is very much worsened and 7 is very much improved since the start of the study.
Time Frame: Week 4 of the Double-blind Treatment Period
Population: FAS of participants with assessments at the timeframe
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Double-blind Treatment Period) | Hydrocodone ER (Double-blind Treatment Period)
Number analyzed (Participants) | 110 | 105
Participants
  General Activities: Very much worsened | 0 | 0
  General Activities: Much worsened | 1 | 1
  General Activities: Slightly worsened | 8 | 3
  General Activities: Unchanged | 31 | 23
  General Activities: Slightly improved | 33 | 38
  General Activities: Much improved | 31 | 29
  General Activities: Very much improved | 6 | 11
  Walking ability: Very much worsened | 0 | 1
  Walking ability: Much worsened | 0 | 0
  Walking ability: Slightly worsened | 8 | 3
  Walking ability: Unchanged | 35 | 27
  Walking ability: Slightly improved | 36 | 36
  Walking ability: Much improved | 26 | 28
  Walking ability: Very much improved | 5 | 10
  Daily living: Very much worsened | 0 | 0
  Daily living: Much worsened | 0 | 2
  Daily living: Slightly worsened | 6 | 3
  Daily living: Unchanged | 36 | 24
  Daily living: Slightly improved | 32 | 39
  Daily living: Much improved | 29 | 29
  Daily living: Very much improved | 7 | 8
  Relationships: Very much worsened | 0 | 0
  Relationships: Much worsened | 0 | 1
  Relationships: Slightly worsened | 3 | 1
  Relationships: Unchanged | 72 | 60
  Relationships: Slightly improved | 13 | 18
  Relationships: Much improved | 16 | 18
  Relationships: Very much improved | 6 | 7
  Enjoyment: Very much worsened | 0 | 1
  Enjoyment: Much worsened | 0 | 0
  Enjoyment: Slightly worsened | 8 | 2
  Enjoyment: Unchanged | 48 | 39
  Enjoyment: Slightly improved | 26 | 26
  Enjoyment: Much improved | 19 | 28
  Enjoyment: Very much improved | 9 | 9

9. Secondary Outcome: Clinician Assessment of Patient Function (CAPF) at Week 8
Description: as for outcome 8
Time Frame: Week 8 of the Double-blind Treatment Period
Population: FAS of participants with assessments at the timeframe
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Double-blind Treatment Period) | Hydrocodone ER (Double-blind Treatment Period)
Number analyzed (Participants) | 98 | 91
Participants
  General Activities: Very much worsened | 0 | 1
  General Activities: Much worsened | 1 | 1
  General Activities: Slightly worsened | 6 | 2
  General Activities: Unchanged | 34 | 23
  General Activities: Slightly improved | 21 | 24
  General Activities: Much improved | 27 | 32
  General Activities: Very much improved | 9 | 8
  Walking ability: Very much worsened | 0 | 1
  Walking ability: Much worsened | 2 | 1
  Walking ability: Slightly worsened | 5 | 1
  Walking ability: Unchanged | 41 | 30
  Walking ability: Slightly improved | 19 | 26
  Walking ability: Much improved | 24 | 26
  Walking ability: Very much improved | 7 | 6
  Daily living: Very much worsened | 0 | 2
  Daily living: Much worsened | 1 | 1
  Daily living: Slightly worsened | 7 | 0
  Daily living: Unchanged | 38 | 25
  Daily living: Slightly improved | 22 | 35
  Daily living: Much improved | 24 | 21
  Daily living: Very much improved | 6 | 7
  Relationships: Very much worsened | 0 | 0
  Relationships: Much worsened | 0 | 0
  Relationships: Slightly worsened | 1 | 2
  Relationships: Unchanged | 68 | 49
  Relationships: Slightly improved | 12 | 19
  Relationships: Much improved | 16 | 17
  Relationships: Very much improved | 3 | 4
  Enjoyment: Very much worsened | 1 | 0
  Enjoyment: Much worsened | 0 | 0
  Enjoyment: Slightly worsened | 7 | 1
  Enjoyment: Unchanged | 38 | 38
  Enjoyment: Slightly improved | 19 | 20
  Enjoyment: Much improved | 27 | 25
  Enjoyment: Very much improved | 6 | 7

10. Secondary Outcome: Clinician Assessment of Patient Function (CAPF) at Week 12
Description: as for outcome 8
Time Frame: Week 12 of the Double-blind Treatment Period
Population: FAS of participants with assessments at the timeframe
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Double-blind Treatment Period) | Hydrocodone ER (Double-blind Treatment Period)
Number analyzed (Participants) | 92 | 86
Participants
  General Activities: Very much worsened | 0 | 0
  General Activities: Much worsened | 0 | 3
  General Activities: Slightly worsened | 4 | 2
  General Activities: Unchanged | 29 | 20
  General Activities: Slightly improved | 29 | 27
  General Activities: Much improved | 19 | 27
  General Activities: Very much improved | 11 | 7
  Walking ability: Very much worsened | 0 | 1
  Walking ability: Much worsened | 0 | 2
  Walking ability: Slightly worsened | 3 | 3
  Walking ability: Unchanged | 38 | 24
  Walking ability: Slightly improved | 26 | 24
  Walking ability: Much improved | 18 | 27
  Walking ability: Very much improved | 7 | 5
  Daily living: Very much worsened | 0 | 0
  Daily living: Much worsened | 0 | 3
  Daily living: Slightly worsened | 6 | 1
  Daily living: Unchanged | 30 | 28
  Daily living: Slightly improved | 26 | 22
  Daily living: Much improved | 20 | 26
  Daily living: Very much improved | 10 | 6
  Relationships: Very much worsened | 0 | 0
  Relationships: Much worsened | 0 | 0
  Relationships: Slightly worsened | 1 | 1
  Relationships: Unchanged | 59 | 47
  Relationships: Slightly improved | 13 | 18
  Relationships: Much improved | 15 | 14
  Relationships: Very much improved | 4 | 6
  Enjoyment: Very much worsened | 0 | 0
  Enjoyment: Much worsened | 0 | 2
  Enjoyment: Slightly worsened | 5 | 3
  Enjoyment: Unchanged | 42 | 31
  Enjoyment: Slightly improved | 16 | 23
  Enjoyment: Much improved | 21 | 21
  Enjoyment: Very much improved | 8 | 6

11. Secondary Outcome: Clinician Assessment of Patient Function (CAPF) at Endpoint
Description: Clinicians assessed participants across 5 dimensions:
  * Patients general activities
  * Patients walking ability
  * Patients ability to work/perform activities of daily living
  * Patients relationships with others
  * Patients enjoyment of life
  Assessments are rated on a 7-point scale, in which 1 is very much worsened and 7 is very much improved since the start of the study.
  Endpoint values are the last observed postbaseline data.
Time Frame: Endpoint of the Double-blind Treatment Period (up to week 12)
Population: FAS of participants with assessments at the timeframe
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Double-blind Treatment Period) | Hydrocodone ER (Double-blind Treatment Period)
Number analyzed (Participants) | 131 | 132
Participants
  General Activities: Very much worsened | 1 | 0
  General Activities: Much worsened | 4 | 5
  General Activities: Slightly worsened | 9 | 4
  General Activities: Unchanged | 46 | 38
  General Activities: Slightly improved | 36 | 37
  General Activities: Much improved | 24 | 40
  General Activities: Very much improved | 11 | 8
  Walking ability: Very much worsened | 1 | 1
  Walking ability: Much worsened | 2 | 4
  Walking ability: Slightly worsened | 7 | 5
  Walking ability: Unchanged | 59 | 45
  Walking ability: Slightly improved | 34 | 32
  Walking ability: Much improved | 21 | 19
  Walking ability: Very much improved | 7 | 6
  Daily living: Very much worsened | 1 | 0
  Daily living: Much worsened | 4 | 6
  Daily living: Slightly worsened | 10 | 3
  Daily living: Unchanged | 49 | 46
  Daily living: Slightly improved | 33 | 33
  Daily living: Much improved | 24 | 36
  Daily living: Very much improved | 10 | 8
  Relationships: Very much worsened | 0 | 0
  Relationships: Much worsened | 1 | 2
  Relationships: Slightly worsened | 3 | 4
  Relationships: Unchanged | 90 | 78
  Relationships: Slightly improved | 15 | 26
  Relationships: Much improved | 18 | 15
  Relationships: Very much improved | 4 | 7
  Enjoyment: Very much worsened | 1 | 0
  Enjoyment: Much worsened | 2 | 5
  Enjoyment: Slightly worsened | 9 | 5
  Enjoyment: Unchanged | 66 | 57
  Enjoyment: Slightly improved | 20 | 31
  Enjoyment: Much improved | 25 | 27
  Enjoyment: Very much improved | 8 | 7

12. Secondary Outcome: Patient Assessment of Function (PAF) at Week 4
Description: The PAF is a self-administered questionnaire used to measure patients' assessment of their own ability to function in normal activities. Answers to the 7 questions were rated on a 7 point scale in which 1 was very much worsened and 7 were very much improved since the start of the study.
  The seven functional areas are:
  * ability to go to work
  * ability to perform at work (includes both work outside the home and housework)
  * ability to walk
  * ability to exercise
  * ability to participate in social events
  * ability to have sex
  * ability to enjoy life
Time Frame: Week 4 of the Double-blind Treatment Period
Population: Full analysis set. Participants contributing to each time point are included in the number analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Double-blind Treatment Period) | Hydrocodone ER (Double-blind Treatment Period)
Number analyzed (Participants) | 147 | 146
Participants
  Go to Work: Very much worsened: number analyzed (Participants) | 75 | 73
  Go to Work: Very much worsened | 0 | 1
  Go to Work: Much worsened: number analyzed (Participants) | 75 | 73
  Go to Work: Much worsened | 2 | 2
  Go to Work: Slightly worsened: number analyzed (Participants) | 75 | 73
  Go to Work: Slightly worsened | 8 | 1
  Go to Work: Unchanged: number analyzed (Participants) | 75 | 73
  Go to Work: Unchanged | 34 | 25
  Go to Work: Slightly improved: number analyzed (Participants) | 75 | 73
  Go to Work: Slightly improved | 13 | 17
  Go to Work: Much improved: number analyzed (Participants) | 75 | 73
  Go to Work: Much improved | 12 | 19
  Go to Work: Very much improved: number analyzed (Participants) | 75 | 73
  Go to Work: Very much improved | 6 | 8
  Perform Work: Very much worsened: number analyzed (Participants) | 108 | 103
  Perform Work: Very much worsened | 0 | 1
  Perform Work: Much worsened: number analyzed (Participants) | 108 | 103
  Perform Work: Much worsened | 3 | 4
  Perform Work: Slightly worsened: number analyzed (Participants) | 108 | 103
  Perform Work: Slightly worsened | 11 | 0
  Perform Work: Unchanged: number analyzed (Participants) | 108 | 103
  Perform Work: Unchanged | 33 | 20
  Perform Work: Slightly improved: number analyzed (Participants) | 108 | 103
  Perform Work: Slightly improved | 32 | 38
  Perform Work: Much improved: number analyzed (Participants) | 108 | 103
  Perform Work: Much improved | 22 | 31
  Perform Work: Very much improved: number analyzed (Participants) | 108 | 103
  Perform Work: Very much improved | 7 | 9
  Walk: Very much worsened: number analyzed (Participants) | 109 | 104
  Walk: Very much worsened | 0 | 0
  Walk: Much worsened: number analyzed (Participants) | 109 | 104
  Walk: Much worsened | 0 | 1
  Walk: Slightly worsened: number analyzed (Participants) | 109 | 104
  Walk: Slightly worsened | 7 | 5
  Walk: Unchanged: number analyzed (Participants) | 109 | 104
  Walk: Unchanged | 37 | 24
  Walk: Slightly improved: number analyzed (Participants) | 109 | 104
  Walk: Slightly improved | 32 | 34
  Walk: Much improved: number analyzed (Participants) | 109 | 104
  Walk: Much improved | 27 | 30
  Walk: Very much improved: number analyzed (Participants) | 109 | 104
  Walk: Very much improved | 6 | 10
  Exercise: Very much worsened: number analyzed (Participants) | 109 | 104
  Exercise: Very much worsened | 1 | 2
  Exercise: Much worsened: number analyzed (Participants) | 109 | 104
  Exercise: Much worsened | 4 | 2
  Exercise: Slightly worsened: number analyzed (Participants) | 109 | 104
  Exercise: Slightly worsened | 6 | 2
  Exercise: Unchanged: number analyzed (Participants) | 109 | 104
  Exercise: Unchanged | 46 | 31
  Exercise: Slightly improved: number analyzed (Participants) | 109 | 104
  Exercise: Slightly improved | 30 | 39
  Exercise: Much improved: number analyzed (Participants) | 109 | 104
  Exercise: Much improved | 18 | 20
  Exercise: Very much improved: number analyzed (Participants) | 109 | 104
  Exercise: Very much improved | 4 | 8
  Social events: Very much worsened: number analyzed (Participants) | 109 | 104
  Social events: Very much worsened | 1 | 0
  Social events: Much worsened: number analyzed (Participants) | 109 | 104
  Social events: Much worsened | 0 | 1
  Social events: Slightly worsened: number analyzed (Participants) | 109 | 104
  Social events: Slightly worsened | 8 | 3
  Social events: Unchanged: number analyzed (Participants) | 109 | 104
  Social events: Unchanged | 52 | 37
  Social events: Slightly improved: number analyzed (Participants) | 109 | 104
  Social events: Slightly improved | 26 | 28
  Social events: Much improved: number analyzed (Participants) | 109 | 104
  Social events: Much improved | 14 | 22
  Social events: Very much improved: number analyzed (Participants) | 109 | 104
  Social events: Very much improved | 8 | 13
  Sex: Very much worsened: number analyzed (Participants) | 107 | 101
  Sex: Very much worsened | 1 | 2
  Sex: Much worsened: number analyzed (Participants) | 107 | 101
  Sex: Much worsened | 5 | 2
  Sex: Slightly worsened: number analyzed (Participants) | 107 | 101
  Sex: Slightly worsened | 8 | 4
  Sex: Unchanged: number analyzed (Participants) | 107 | 101
  Sex: Unchanged | 66 | 64
  Sex: Slightly improved: number analyzed (Participants) | 107 | 101
  Sex: Slightly improved | 18 | 7
  Sex: Much improved: number analyzed (Participants) | 107 | 101
  Sex: Much improved | 5 | 15
  Sex: Very much improved: number analyzed (Participants) | 107 | 101
  Sex: Very much improved | 4 | 7
  Enjoy life: Very much worsened: number analyzed (Participants) | 109 | 104
  Enjoy life: Very much worsened | 1 | 0
  Enjoy life: Much worsened: number analyzed (Participants) | 109 | 104
  Enjoy life: Much worsened | 0 | 2
  Enjoy life: Slightly worsened: number analyzed (Participants) | 109 | 104
  Enjoy life: Slightly worsened | 8 | 4
  Enjoy life: Unchanged: number analyzed (Participants) | 109 | 104
  Enjoy life: Unchanged | 41 | 34
  Enjoy life: Slightly improved: number analyzed (Participants) | 109 | 104
  Enjoy life: Slightly improved | 28 | 27
  Enjoy life: Much improved: number analyzed (Participants) | 109 | 104
  Enjoy life: Much improved | 20 | 28
  Enjoy life: Very much improved: number analyzed (Participants) | 109 | 104
  Enjoy life: Very much improved | 11 | 9

13. Secondary Outcome: Patient Assessment of Function (PAF) at Week 8
Description: as for outcome 12
Time Frame: Week 8 of the Double-blind Treatment Period
Population: Full analysis set. Participants contributing to each time point are included in the number analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Double-blind Treatment Period) | Hydrocodone ER (Double-blind Treatment Period)
Number analyzed (Participants) | 147 | 146
Participants
  Go to Work: Very much worsened: number analyzed (Participants) | 65 | 64
  Go to Work: Very much worsened | 0 | 2
  Go to Work: Much worsened: number analyzed (Participants) | 65 | 64
  Go to Work: Much worsened | 0 | 0
  Go to Work: Slightly worsened: number analyzed (Participants) | 65 | 64
  Go to Work: Slightly worsened | 7 | 3
  Go to Work: Unchanged: number analyzed (Participants) | 65 | 64
  Go to Work: Unchanged | 31 | 29
  Go to Work: Slightly improved: number analyzed (Participants) | 65 | 64
  Go to Work: Slightly improved | 10 | 9
  Go to Work: Much improved: number analyzed (Participants) | 65 | 64
  Go to Work: Much improved | 14 | 18
  Go to Work: Very much improved: number analyzed (Participants) | 65 | 64
  Go to Work: Very much improved | 3 | 3
  Perform Work: Very much worsened: number analyzed (Participants) | 97 | 93
  Perform Work: Very much worsened | 1 | 2
  Perform Work: Much worsened: number analyzed (Participants) | 97 | 93
  Perform Work: Much worsened | 3 | 0
  Perform Work: Slightly worsened: number analyzed (Participants) | 97 | 93
  Perform Work: Slightly worsened | 7 | 6
  Perform Work: Unchanged: number analyzed (Participants) | 97 | 93
  Perform Work: Unchanged | 38 | 22
  Perform Work: Slightly improved: number analyzed (Participants) | 97 | 93
  Perform Work: Slightly improved | 22 | 25
  Perform Work: Much improved: number analyzed (Participants) | 97 | 93
  Perform Work: Much improved | 17 | 33
  Perform Work: Very much improved: number analyzed (Participants) | 97 | 93
  Perform Work: Very much improved | 9 | 5
  Walk: Very much worsened: number analyzed (Participants) | 98 | 93
  Walk: Very much worsened | 0 | 1
  Walk: Much worsened: number analyzed (Participants) | 98 | 93
  Walk: Much worsened | 2 | 2
  Walk: Slightly worsened: number analyzed (Participants) | 98 | 93
  Walk: Slightly worsened | 7 | 4
  Walk: Unchanged: number analyzed (Participants) | 98 | 93
  Walk: Unchanged | 40 | 22
  Walk: Slightly improved: number analyzed (Participants) | 98 | 93
  Walk: Slightly improved | 23 | 27
  Walk: Much improved: number analyzed (Participants) | 98 | 93
  Walk: Much improved | 17 | 27
  Walk: Very much improved: number analyzed (Participants) | 98 | 93
  Walk: Very much improved | 9 | 10
  Exercise: Very much worsened: number analyzed (Participants) | 98 | 93
  Exercise: Very much worsened | 0 | 2
  Exercise: Much worsened: number analyzed (Participants) | 98 | 93
  Exercise: Much worsened | 3 | 1
  Exercise: Slightly worsened: number analyzed (Participants) | 98 | 93
  Exercise: Slightly worsened | 8 | 8
  Exercise: Unchanged: number analyzed (Participants) | 98 | 93
  Exercise: Unchanged | 42 | 28
  Exercise: Slightly improved: number analyzed (Participants) | 98 | 93
  Exercise: Slightly improved | 23 | 28
  Exercise: Much improved: number analyzed (Participants) | 98 | 93
  Exercise: Much improved | 16 | 21
  Exercise: Very much improved: number analyzed (Participants) | 98 | 93
  Exercise: Very much improved | 6 | 5
  Social events: Very much worsened: number analyzed (Participants) | 98 | 93
  Social events: Very much worsened | 1 | 0
  Social events: Much worsened: number analyzed (Participants) | 98 | 93
  Social events: Much worsened | 1 | 2
  Social events: Slightly worsened: number analyzed (Participants) | 98 | 93
  Social events: Slightly worsened | 3 | 2
  Social events: Unchanged: number analyzed (Participants) | 98 | 93
  Social events: Unchanged | 48 | 42
  Social events: Slightly improved: number analyzed (Participants) | 98 | 93
  Social events: Slightly improved | 18 | 19
  Social events: Much improved: number analyzed (Participants) | 98 | 93
  Social events: Much improved | 18 | 19
  Social events: Very much improved: number analyzed (Participants) | 98 | 93
  Social events: Very much improved | 9 | 9
  Sex: Very much worsened: number analyzed (Participants) | 95 | 91
  Sex: Very much worsened | 0 | 1
  Sex: Much worsened: number analyzed (Participants) | 95 | 91
  Sex: Much worsened | 1 | 0
  Sex: Slightly worsened: number analyzed (Participants) | 95 | 91
  Sex: Slightly worsened | 3 | 9
  Sex: Unchanged: number analyzed (Participants) | 95 | 91
  Sex: Unchanged | 74 | 52
  Sex: Slightly improved: number analyzed (Participants) | 95 | 91
  Sex: Slightly improved | 9 | 12
  Sex: Much improved: number analyzed (Participants) | 95 | 91
  Sex: Much improved | 4 | 14
  Sex: Very much improved: number analyzed (Participants) | 95 | 91
  Sex: Very much improved | 4 | 3
  Enjoy life: Very much worsened: number analyzed (Participants) | 98 | 93
  Enjoy life: Very much worsened | 1 | 0
  Enjoy life: Much worsened: number analyzed (Participants) | 98 | 93
  Enjoy life: Much worsened | 1 | 1
  Enjoy life: Slightly worsened: number analyzed (Participants) | 98 | 93
  Enjoy life: Slightly worsened | 6 | 3
  Enjoy life: Unchanged: number analyzed (Participants) | 98 | 93
  Enjoy life: Unchanged | 41 | 34
  Enjoy life: Slightly improved: number analyzed (Participants) | 98 | 93
  Enjoy life: Slightly improved | 24 | 25
  Enjoy life: Much improved: number analyzed (Participants) | 98 | 93
  Enjoy life: Much improved | 23 | 23
  Enjoy life: Very much improved: number analyzed (Participants) | 98 | 93
  Enjoy life: Very much improved | 3 | 7

14. Secondary Outcome: Patient Assessment of Function (PAF) at Week 12
Description: as for outcome 12
Time Frame: Week 12 of the Double-blind Treatment Period
Population: Full analysis set. Participants contributing to each time point are included in the number analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Double-blind Treatment Period) | Hydrocodone ER (Double-blind Treatment Period)
Number analyzed (Participants) | 147 | 146
Participants
  Go to Work: Very much worsened: number analyzed (Participants) | 60 | 61
  Go to Work: Very much worsened | 0 | 1
  Go to Work: Much worsened: number analyzed (Participants) | 60 | 61
  Go to Work: Much worsened | 2 | 1
  Go to Work: Slightly worsened: number analyzed (Participants) | 60 | 61
  Go to Work: Slightly worsened | 5 | 3
  Go to Work: Unchanged: number analyzed (Participants) | 60 | 61
  Go to Work: Unchanged | 27 | 19
  Go to Work: Slightly improved: number analyzed (Participants) | 60 | 61
  Go to Work: Slightly improved | 7 | 18
  Go to Work: Much improved: number analyzed (Participants) | 60 | 61
  Go to Work: Much improved | 13 | 17
  Go to Work: Very much improved: number analyzed (Participants) | 60 | 61
  Go to Work: Very much improved | 6 | 2
  Perform Work: Very much worsened: number analyzed (Participants) | 91 | 84
  Perform Work: Very much worsened | 1 | 1
  Perform Work: Much worsened: number analyzed (Participants) | 91 | 84
  Perform Work: Much worsened | 0 | 3
  Perform Work: Slightly worsened: number analyzed (Participants) | 91 | 84
  Perform Work: Slightly worsened | 10 | 5
  Perform Work: Unchanged: number analyzed (Participants) | 91 | 84
  Perform Work: Unchanged | 26 | 20
  Perform Work: Slightly improved: number analyzed (Participants) | 91 | 84
  Perform Work: Slightly improved | 26 | 26
  Perform Work: Much improved: number analyzed (Participants) | 91 | 84
  Perform Work: Much improved | 21 | 25
  Perform Work: Very much improved: number analyzed (Participants) | 91 | 84
  Perform Work: Very much improved | 7 | 4
  Walk: Very much worsened: number analyzed (Participants) | 91 | 85
  Walk: Very much worsened | 1 | 1
  Walk: Much worsened: number analyzed (Participants) | 91 | 85
  Walk: Much worsened | 2 | 2
  Walk: Slightly worsened: number analyzed (Participants) | 91 | 85
  Walk: Slightly worsened | 10 | 5
  Walk: Unchanged: number analyzed (Participants) | 91 | 85
  Walk: Unchanged | 29 | 20
  Walk: Slightly improved: number analyzed (Participants) | 91 | 85
  Walk: Slightly improved | 20 | 27
  Walk: Much improved: number analyzed (Participants) | 91 | 85
  Walk: Much improved | 23 | 23
  Walk: Very much improved: number analyzed (Participants) | 91 | 85
  Walk: Very much improved | 6 | 7
  Exercise: Very much worsened: number analyzed (Participants) | 91 | 85
  Exercise: Very much worsened | 2 | 1
  Exercise: Much worsened: number analyzed (Participants) | 91 | 85
  Exercise: Much worsened | 2 | 3
  Exercise: Slightly worsened: number analyzed (Participants) | 91 | 85
  Exercise: Slightly worsened | 9 | 4
  Exercise: Unchanged: number analyzed (Participants) | 91 | 85
  Exercise: Unchanged | 34 | 30
  Exercise: Slightly improved: number analyzed (Participants) | 91 | 85
  Exercise: Slightly improved | 23 | 26
  Exercise: Much improved: number analyzed (Participants) | 91 | 85
  Exercise: Much improved | 15 | 14
  Exercise: Very much improved: number analyzed (Participants) | 91 | 85
  Exercise: Very much improved | 6 | 7
  Social events: Very much worsened: number analyzed (Participants) | 91 | 85
  Social events: Very much worsened | 1 | 0
  Social events: Much worsened: number analyzed (Participants) | 91 | 85
  Social events: Much worsened | 0 | 2
  Social events: Slightly worsened: number analyzed (Participants) | 91 | 85
  Social events: Slightly worsened | 7 | 6
  Social events: Unchanged: number analyzed (Participants) | 91 | 85
  Social events: Unchanged | 45 | 29
  Social events: Slightly improved: number analyzed (Participants) | 91 | 85
  Social events: Slightly improved | 16 | 25
  Social events: Much improved: number analyzed (Participants) | 91 | 85
  Social events: Much improved | 17 | 16
  Social events: Very much improved: number analyzed (Participants) | 91 | 85
  Social events: Very much improved | 5 | 7
  Sex: Very much worsened: number analyzed (Participants) | 91 | 82
  Sex: Very much worsened | 2 | 0
  Sex: Much worsened: number analyzed (Participants) | 91 | 82
  Sex: Much worsened | 2 | 4
  Sex: Slightly worsened: number analyzed (Participants) | 91 | 82
  Sex: Slightly worsened | 7 | 7
  Sex: Unchanged: number analyzed (Participants) | 91 | 82
  Sex: Unchanged | 64 | 46
  Sex: Slightly improved: number analyzed (Participants) | 91 | 82
  Sex: Slightly improved | 7 | 11
  Sex: Much improved: number analyzed (Participants) | 91 | 82
  Sex: Much improved | 6 | 12
  Sex: Very much improved: number analyzed (Participants) | 91 | 82
  Sex: Very much improved | 3 | 2
  Enjoy life: Very much worsened: number analyzed (Participants) | 91 | 85
  Enjoy life: Very much worsened | 1 | 0
  Enjoy life: Much worsened: number analyzed (Participants) | 91 | 85
  Enjoy life: Much worsened | 0 | 4
  Enjoy life: Slightly worsened: number analyzed (Participants) | 91 | 85
  Enjoy life: Slightly worsened | 7 | 4
  Enjoy life: Unchanged: number analyzed (Participants) | 91 | 85
  Enjoy life: Unchanged | 36 | 27
  Enjoy life: Slightly improved: number analyzed (Participants) | 91 | 85
  Enjoy life: Slightly improved | 21 | 18
  Enjoy life: Much improved: number analyzed (Participants) | 91 | 85
  Enjoy life: Much improved | 18 | 24
  Enjoy life: Very much improved: number analyzed (Participants) | 91 | 85
  Enjoy life: Very much improved | 8 | 8

15. Secondary Outcome: Patient Assessment of Function (PAF) at Endpoint
Description: The PAF is a self-administered questionnaire used to measure patients' assessment of their own ability to function in normal activities. Answers to the 7 questions were rated on a 7 point scale in which 1 was very much worsened and 7 were very much improved since the start of the study.
  The seven functional areas are:
  * ability to go to work
  * ability to perform at work (includes both work outside the home and housework)
  * ability to walk
  * ability to exercise
  * ability to participate in social events
  * ability to have sex
  * ability to enjoy life
  Endpoint values are the last observed postbaseline data.
Time Frame: Endpoint of the Double-blind Treatment Period (up to week 12)
Population: Full analysis set. Participants contributing to each time point are included in the number analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Double-blind Treatment Period) | Hydrocodone ER (Double-blind Treatment Period)
Number analyzed (Participants) | 147 | 146
Participants
  Go to Work: Very much worsened: number analyzed (Participants) | 99 | 106
  Go to Work: Very much worsened | 0 | 1
  Go to Work: Much worsened: number analyzed (Participants) | 99 | 106
  Go to Work: Much worsened | 4 | 2
  Go to Work: Slightly worsened: number analyzed (Participants) | 99 | 106
  Go to Work: Slightly worsened | 10 | 6
  Go to Work: Unchanged: number analyzed (Participants) | 99 | 106
  Go to Work: Unchanged | 47 | 39
  Go to Work: Slightly improved: number analyzed (Participants) | 99 | 106
  Go to Work: Slightly improved | 11 | 26
  Go to Work: Much improved: number analyzed (Participants) | 99 | 106
  Go to Work: Much improved | 21 | 26
  Go to Work: Very much improved: number analyzed (Participants) | 99 | 106
  Go to Work: Very much improved | 6 | 6
  Perform Work: Very much worsened: number analyzed (Participants) | 131 | 133
  Perform Work: Very much worsened | 2 | 2
  Perform Work: Much worsened: number analyzed (Participants) | 131 | 133
  Perform Work: Much worsened | 3 | 5
  Perform Work: Slightly worsened: number analyzed (Participants) | 131 | 133
  Perform Work: Slightly worsened | 17 | 12
  Perform Work: Unchanged: number analyzed (Participants) | 131 | 133
  Perform Work: Unchanged | 43 | 34
  Perform Work: Slightly improved: number analyzed (Participants) | 131 | 133
  Perform Work: Slightly improved | 31 | 39
  Perform Work: Much improved: number analyzed (Participants) | 131 | 133
  Perform Work: Much improved | 27 | 34
  Perform Work: Very much improved: number analyzed (Participants) | 131 | 133
  Perform Work: Very much improved | 8 | 7
  Walk: Very much worsened: number analyzed (Participants) | 131 | 133
  Walk: Very much worsened | 1 | 1
  Walk: Much worsened: number analyzed (Participants) | 131 | 133
  Walk: Much worsened | 7 | 4
  Walk: Slightly worsened: number analyzed (Participants) | 131 | 133
  Walk: Slightly worsened | 13 | 10
  Walk: Unchanged: number analyzed (Participants) | 131 | 133
  Walk: Unchanged | 47 | 36
  Walk: Slightly improved: number analyzed (Participants) | 131 | 133
  Walk: Slightly improved | 28 | 40
  Walk: Much improved: number analyzed (Participants) | 131 | 133
  Walk: Much improved | 28 | 32
  Walk: Very much improved: number analyzed (Participants) | 131 | 133
  Walk: Very much improved | 7 | 10
  Exercise: Very much worsened: number analyzed (Participants) | 131 | 133
  Exercise: Very much worsened | 4 | 3
  Exercise: Much worsened: number analyzed (Participants) | 131 | 133
  Exercise: Much worsened | 6 | 5
  Exercise: Slightly worsened: number analyzed (Participants) | 131 | 133
  Exercise: Slightly worsened | 13 | 9
  Exercise: Unchanged: number analyzed (Participants) | 131 | 133
  Exercise: Unchanged | 52 | 51
  Exercise: Slightly improved: number analyzed (Participants) | 131 | 133
  Exercise: Slightly improved | 30 | 30
  Exercise: Much improved: number analyzed (Participants) | 131 | 133
  Exercise: Much improved | 19 | 24
  Exercise: Very much improved: number analyzed (Participants) | 131 | 133
  Exercise: Very much improved | 7 | 9
  Social events: Very much worsened: number analyzed (Participants) | 131 | 133
  Social events: Very much worsened | 1 | 1
  Social events: Much worsened: number analyzed (Participants) | 131 | 133
  Social events: Much worsened | 3 | 4
  Social events: Slightly worsened: number analyzed (Participants) | 131 | 133
  Social events: Slightly worsened | 10 | 12
  Social events: Unchanged: number analyzed (Participants) | 131 | 133
  Social events: Unchanged | 67 | 51
  Social events: Slightly improved: number analyzed (Participants) | 131 | 133
  Social events: Slightly improved | 23 | 30
  Social events: Much improved: number analyzed (Participants) | 131 | 133
  Social events: Much improved | 21 | 25
  Social events: Very much improved: number analyzed (Participants) | 131 | 133
  Social events: Very much improved | 6 | 10
  Sex: Very much worsened: number analyzed (Participants) | 131 | 129
  Sex: Very much worsened | 3 | 0
  Sex: Much worsened: number analyzed (Participants) | 131 | 129
  Sex: Much worsened | 6 | 6
  Sex: Slightly worsened: number analyzed (Participants) | 131 | 129
  Sex: Slightly worsened | 10 | 12
  Sex: Unchanged: number analyzed (Participants) | 131 | 129
  Sex: Unchanged | 88 | 76
  Sex: Slightly improved: number analyzed (Participants) | 131 | 129
  Sex: Slightly improved | 12 | 13
  Sex: Much improved: number analyzed (Participants) | 131 | 129
  Sex: Much improved | 8 | 18
  Sex: Very much improved: number analyzed (Participants) | 131 | 129
  Sex: Very much improved | 4 | 4
  Enjoy life: Very much worsened: number analyzed (Participants) | 131 | 132
  Enjoy life: Very much worsened | 2 | 0
  Enjoy life: Much worsened: number analyzed (Participants) | 131 | 132
  Enjoy life: Much worsened | 3 | 7
  Enjoy life: Slightly worsened: number analyzed (Participants) | 131 | 132
  Enjoy life: Slightly worsened | 10 | 9
  Enjoy life: Unchanged: number analyzed (Participants) | 131 | 132
  Enjoy life: Unchanged | 59 | 45
  Enjoy life: Slightly improved: number analyzed (Participants) | 131 | 132
  Enjoy life: Slightly improved | 27 | 25
  Enjoy life: Much improved: number analyzed (Participants) | 131 | 132
  Enjoy life: Much improved | 21 | 35
  Enjoy life: Very much improved: number analyzed (Participants) | 131 | 132
  Enjoy life: Very much improved | 9 | 11

16. Secondary Outcome: Clinician Global Impression of Severity (CGI-S) of Illness Scores During the Double-blind Treatment Period
Description: The CGI-S is a clinician-rated scale that assesses the severity of the patient's pain condition and response to the treatment. Severity of illness, as related to moderate to severe pain, consists of the following 7 categories:
  * 1 normal-shows no sign of illness,
  * 2 borderline ill,
  * 3 mildly (slightly) ill,
  * 4 moderately ill,
  * 5 markedly ill,
  * 6 severely ill, and
  * 7 among the most extremely ill (Guy 1976).
  The clinician assesses the severity of the patient's condition, based on the clinician's total clinical experience with patients with this condition, in response to treatment.
  Endpoint values are the last observed postbaseline data.
Time Frame: Baseline (end of Open-Label Titration Period), Weeks 1, 2, 4, 8, and 12 of the Double-blind treatment period
Population: Full analysis set. Participants contributing to each time point are included in the number analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo (Double-blind Treatment Period) | Hydrocodone ER (Double-blind Treatment Period)
Number analyzed (Participants) | 147 | 146
units on a scale
  Baseline | 3.0 (1.19) | 2.8 (1.07)
  Week 1: number analyzed (Participants) | 136 | 132
  Week 1 | 2.9 (1.16) | 2.9 (1.10)
  Week 2: number analyzed (Participants) | 127 | 122
  Week 2 | 2.9 (1.20) | 2.8 (1.07)
  Week 4: number analyzed (Participants) | 110 | 105
  Week 4 | 2.9 (1.26) | 2.7 (1.03)
  Week 8: number analyzed (Participants) | 98 | 93
  Week 8 | 2.8 (1.21) | 2.7 (1.01)
  Week 12: number analyzed (Participants) | 92 | 86
  Week 12 | 2.8 (1.19) | 2.7 (1.08)
  Endpoint: number analyzed (Participants) | 146 | 143
  Endpoint | 2.9 (1.18) | 2.8 (1.12)

17. Secondary Outcome: Short-Form Health Survey (SF-36) Physical and Mental Component Summary Scores at Baseline, Week 12 and Endpoint
Description: SF-36 is a generic 36-item questionnaire measuring health-related quality of life (HRQL) covering 2 summary measures: physical component summary (PCS) and mental component summary (MCS). The SF-36 consists of 8 subscales. The PCS is represented by 4 subscales: physical function, role limitations due to physical problems, pain, and general health perception. The MCS is represented by 4 subscales: vitality, social function, role limitations due to emotional problems, and mental health. Participants self-report on items in a subscale that have between 2-6 choices per item using Likert-type responses (e.g. none of the time, some of the time, etc.). PCS and MCS scores are constructed as a T-score with a mean of 50 and standard deviation of 10 and no minimum or maximum score; higher scores indicate better health status.
Time Frame: Baseline (end of Open-Label Titration Period), Week 12 and Endpoint (last visit up to week 12) of the Double-blind treatment period
Population: Full analysis set. Participants contributing to each time point are included in the number analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo (Double-blind Treatment Period) | Hydrocodone ER (Double-blind Treatment Period)
Number analyzed (Participants) | 147 | 146
units on a scale
  PCS - Baseline | 35.5 (8.96) | 35.8 (9.28)
  PCS - Week 12: number analyzed (Participants) | 93 | 84
  PCS - Week 12 | 36.9 (10.04) | 37.6 (9.04)
  PCS - Endpoint: number analyzed (Participants) | 120 | 122
  PCS - Endpoint | 35.9 (10.13) | 36.9 (9.16)
  MCS - Baseline | 52.8 (9.99) | 52.8 (10.47)
  MCS - Week 12: number analyzed (Participants) | 93 | 84
  MCS - Week 12 | 54.7 (9.71) | 53.6 (8.06)
  MCS - Endpoint: number analyzed (Participants) | 120 | 122
  MCS - Endpoint | 54.0 (10.27) | 52.6 (9.22)

18. Secondary Outcome: Brief Pain Inventory - Short Form (BPI-SF) Pain Interference Mean Score During the Double-Blind Treatment Period
Description: For pain interference, the BPI-SF used numerical scales to measure how much pain had interfered with 7 daily activities, including general activity, walking, work, mood, enjoyment of life, relations with others, and sleep in the past 24 hours. The scale used an 11 point Likert scale; range: 0 [does not interfere] to 10 [completely interferes]. BPI pain interference was typically scored as the mean of the 7 interference items. This mean could be used if at least 4 of 7 items had been completed on a given administration.
Time Frame: Baseline (end of Open-Label Titration Period), Weeks 1, 2, 4, 8, 12 and Endpoint (last visit up to week 12) of the Double-blind treatment period
Population: Full analysis set. Participants contributing to each time point are included in the number analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Hydrocodone ER (Double-blind Treatment Period): Participants were administered ER hydrocodone tablets at a dosage deemed successful for managing their pain during the titration period. Dosages of 15, 30, 45, 60, or 90 mg every 12 hours were given for 12 weeks during the double-blind period.
Arm/Group | Placebo (Double-blind Treatment Period) | Hydrocodone ER (Double-blind Treatment Period)
Number analyzed (Participants) | 147 | 146
units on a scale
  Baseline | 2.9 (2.09) | 2.8 (2.05)
  Week 1: number analyzed (Participants) | 136 | 130
  Week 1 | 3.0 (2.23) | 3.1 (2.22)
  Week 2: number analyzed (Participants) | 130 | 123
  Week 2 | 2.9 (2.25) | 2.7 (2.19)
  Week 4: number analyzed (Participants) | 115 | 111
  Week 4 | 2.9 (2.39) | 2.8 (2.06)
  Week 8: number analyzed (Participants) | 106 | 100
  Week 8 | 2.9 (2.37) | 2.9 (2.23)
  Week 12: number analyzed (Participants) | 102 | 94
  Week 12 | 3.0 (2.31) | 3.3 (2.30)
  Endpoint: number analyzed (Participants) | 146 | 144
  Endpoint | 3.5 (2.45) | 3.3 (2.28)

19. Secondary Outcome: Participants With Adverse Events
Description: An adverse event (AE) was defined in the protocol as any untoward medical occurrence that develops or worsens in severity during the conduct of a clinical study and does not necessarily have a causal relationship to the study drug. Severity was rated by the investigator on a scale of mild, moderate and severe, with severe= an inability to carry out usual activities. Relation of AE to treatment was determined by the investigator. Serious AEs include death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, OR an important medical event that jeopardized the patient and required medical intervention to prevent the previously listed serious outcomes.
Time Frame: Day 1 up to Day 52 in Open-Label Titration; Day 1 up to Day 128 in Double-Blind Treatment period
Population: Safety analysis set (Open-Label Titration) and FAS (Double-Blind Treatment)
Measure: Count of Participants; unit: Participants
Groups:
- Open-Label Titration: Opioid Naive: During the open label titration period, all participants received hydrocodone extended release tablets on an open-label basis. Opioid naïve participants (ie, those taking less than 10 mg/day of oxycodone or equivalent, during the 14 days before screening) started at a 15 mg dose of hydrocodone extended release, administered every 12 hours. A decision regarding dose adjustment was made based on whether the criterion of successful dose (ie, dose that produced stable pain relief) was met. In general, dose escalation stepped from 15 mg to 30 mg, 45 mg, 60 mg, and 90 mg every 12 hours until stable pain relief was obtained.
- Open-Label Titration: Opioid Experienced: During the open label titration period, all participants received hydrocodone extended release tablets on an open-label basis. Opioid experienced participants switched from their current opioid medications to the calculated dose of hydrocodone extended release tablets based on an equianalgesic dose-conversion scheme.
  A decision regarding dose adjustment was made based on whether the criterion of successful dose (ie, dose that produced stable pain relief) was met. In general, dose escalation stepped to 30 mg or 45 mg or 60 mg, or 90 mg every 12 hours until stable pain relief was obtained. The escalated dose was dependent upon the initial calculated equivalent dose.
Arm/Group | Open-Label Titration: Opioid Naive | Open-Label Titration: Opioid Experienced | Placebo (Double-blind Treatment Period) | Hydrocodone ER (Double-blind Treatment Period)
Number analyzed (Participants) | 189 | 200 | 147 | 146
Participants
  Any adverse event | 111 | 116 | 91 | 93
  Severe adverse event | 9 | 8 | 7 | 9
  Treatment-related adverse event | 90 | 72 | 28 | 48
  Deaths | 0 | 0 | 0 | 0
  Serious adverse event | 0 | 2 | 3 | 3
  Withdrawals from treatment due to AE | 33 | 15 | 3 | 9

20. Secondary Outcome: Participants With Potentially Clinically Significant Abnormal Vital Signs Values During the Double-Blind Treatment Period
Description: Data represents participants with potentially clinically significant (PCS) vital sign values.
  Significance criteria
  * Pulse - high: >=120 and increase of >= 15 beats/minute from baseline
  * Pulse - low: <=50 and decrease of >=15 beats/minute
  * Systolic blood pressure - high: >=180 and increase >=20 mmHg
  * Systolic blood pressure - low: <=90 and decrease >=20 mmHg
  * Diastolic blood pressure - high: >=105 and increase of >=15 mmHg
  * Diastolic blood pressure - low: <=50 and decrease of >=15 mmHg
Time Frame: Day 1 up to Day 128 in Double-Blind Treatment period
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Double-blind Treatment Period) | Hydrocodone ER (Double-blind Treatment Period)
Number analyzed (Participants) | 147 | 146
Participants
  At least one clinically significant vital sign | 2 | 5
  Pulse - high | 0 | 0
  Pulse - low | 0 | 0
  Systolic blood pressure - high | 1 | 0
  Systolic blood pressure - low | 1 | 3
  Diastolic blood pressure - high | 0 | 2
  Diastolic blood pressure - low | 0 | 1

21. Secondary Outcome: Participants With Potentially Clinically Significant Abnormal Laboratory Values During the Double-Blind Treatment Period
Description: Data represents participants with potentially clinically significant abnormal serum chemistry, hematology and urinalysis values.
  Significance criteria:
  * Blood urea nitrogen: >=10.71 mmol/L
  * Uric acid: M>=625, F>=506 μmol/L
  * Hemoglobin: M<=115, F<=95 g/dL
  * Hematocrit: M<0.37, F<0.32 %
  * Urinalysis: blood (hemoglobin) and total protein: >=2 unit increase from baseline
Time Frame: Day 1 up to Day 128 in Double-Blind Treatment period
Population: Full analysis set including participants with laboratory assessments
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Double-blind Treatment Period) | Hydrocodone ER (Double-blind Treatment Period)
Number analyzed (Participants) | 147 | 146
Participants
  Blood urea nitrogen: number analyzed (Participants) | 145 | 144
  Blood urea nitrogen | 1 | 4
  Uric acid: number analyzed (Participants) | 145 | 144
  Uric acid | 2 | 5
  Hemoglobin: number analyzed (Participants) | 146 | 143
  Hemoglobin | 1 | 3
  Hematocrit: number analyzed (Participants) | 144 | 141
  Hematocrit | 1 | 5
  Urine blood: number analyzed (Participants) | 146 | 139
  Urine blood | 2 | 3
  Urine total protein: number analyzed (Participants) | 146 | 139
  Urine total protein | 1 | 0

22. Secondary Outcome: Subjective Opiate Withdrawal Scales (SOWS) Scores During the Double-Blind Treatment Period
Description: The results of the SOWS were collected in the e-diary daily during the first 4 weeks of the double blind treatment period and then during clinic visits at weeks 8 and 12 or early termination. The SOWS was a self administered questionnaire used to measure a participant's signs and symptoms of withdrawal from opiates. The scale contained 16 symptoms (eg, my nose is running; I feel restless), the participant rated the intensity on a scale of 0 (not at all) to 4 (extremely) for a total score of 0-64. The daily total score for the first 4 weeks was the largest score observed during the time period preceding that visit. For example, the week 1 score for each participant was the largest total score on any day between baseline and the night before the week 1 visit; the week 4 score for each participant was the largest score observed between the week 2 visit and the night before the week 4 visit.
Time Frame: Weeks 1, 2, 4, 8, 12 and Endpoint (last visit up to Week 12) of the Double-blind treatment period
Population: Full analysis set. Participants contributing to each time point are included in the number analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo (Double-blind Treatment Period) | Hydrocodone ER (Double-blind Treatment Period)
Number analyzed (Participants) | 147 | 146
units on a scale
  Week 1: number analyzed (Participants) | 143 | 142
  Week 1 | 5.9 (5.39) | 6.1 (5.93)
  Week 2: number analyzed (Participants) | 135 | 128
  Week 2 | 5.4 (5.59) | 4.4 (5.10)
  Week 4: number analyzed (Participants) | 130 | 123
  Week 4 | 5.5 (6.16) | 5.3 (5.37)
  Week 8: number analyzed (Participants) | 106 | 99
  Week 8 | 3.4 (4.68) | 3.2 (4.23)
  Week 12: number analyzed (Participants) | 100 | 94
  Week 12 | 3.2 (4.73) | 3.6 (5.29)
  Endpoint | 3.6 (4.96) | 4.3 (6.30)

23. Secondary Outcome: Clinical Opiate Withdrawal Scales (COWS) Scores During the Double-Blind Treatment Period
Description: The COWS was a clinician rated scale used to measure a participant's signs and symptoms of withdrawal from opiates, with ratings based only on apparent relationship to withdrawal. The COWS was performed at day 0 and weeks 1, 2, 4, 8, and 12 (double blind treatment period) or early termination. The scale contained 11 signs/symptoms whose intensity the clinician rated on a scale of 0 to 4 or 5.
  A total score was calculated as the sum of the responses to the 11 signs/symptoms for a total range of 0-48. Withdrawal severity was classified, based on the total score, as follows:
  * 0 to 4=normal
  * 5 to 12=mild
  * 13 to 24=moderate
  * 25 to 36=moderately severe
  * >36=severe
Time Frame: as for outcome 18
Population: Full analysis set. Participants contributing to each time point are included in the number analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo (Double-blind Treatment Period) | Hydrocodone ER (Double-blind Treatment Period)
Number analyzed (Participants) | 147 | 146
units on a scale
  Baseline: number analyzed (Participants) | 146 | 146
  Baseline | 0.5 (0.90) | 0.5 (0.90)
  Week 1: number analyzed (Participants) | 136 | 132
  Week 1 | 0.8 (1.51) | 0.7 (1.29)
  Week 2: number analyzed (Participants) | 130 | 123
  Week 2 | 0.7 (1.33) | 0.5 (0.92)
  Week 4: number analyzed (Participants) | 116 | 111
  Week 4 | 0.8 (1.58) | 0.6 (1.22)
  Week 8: number analyzed (Participants) | 106 | 100
  Week 8 | 0.7 (1.34) | 0.6 (1.15)
  Week 12: number analyzed (Participants) | 101 | 94
  Week 12 | 0.5 (0.92) | 0.8 (1.76)
  Endpoint | 0.7 (1.13) | 1.1 (2.02)

24. Secondary Outcome: Addiction Behavior Checklist (ABC) Total Scores During Both the Open-Label Titration and Double-Blind Treatment Periods
Description: The ABC was a clinician rated scale that consisted of a brief (20 item) questionnaire designed to track behaviors characteristic of addiction related to prescription opioid medications in chronic pain populations. Items were focused on observable behaviors noted both during and between clinic visits. Each affirmative response was counted as one point, and points were added to calculate the total score, consequently resulting in scores ranging from 0 to 20 (0=no addiction-related behaviors seen and higher scores indicating an increasing number of addition-related behaviors seen).
  The ABC was to be performed at visits 2 and 7 (beginning and end of Open-label Titration period) and weeks 1, 4, 8, and 12 (Double-blind Treatment period) or early termination.
Time Frame: Baseline for Open-Label Titration period, Baseline for Double-Blind Treatment period (which is also the end of the Open-Label Titration period), Weeks 1, 4, 8, 12, and Endpoint (last visit up to Week 12) of the Double-blind Treatment period
Population: Full analysis set. Participants contributing to each time point are included in the number analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo (Double-blind Treatment Period) | Hydrocodone ER (Double-blind Treatment Period)
Number analyzed (Participants) | 147 | 146
units on a scale
  Baseline Open-Label Titration: number analyzed (Participants) | 146 | 143
  Baseline Open-Label Titration | 0.3 (0.65) | 0.3 (0.70)
  Baseline Double-blind Treatment | 0.1 (0.39) | 0.2 (0.43)
  Week 1: number analyzed (Participants) | 136 | 132
  Week 1 | 0.2 (0.47) | 0.2 (0.50)
  Week 4: number analyzed (Participants) | 116 | 111
  Week 4 | 0.1 (0.40) | 0.3 (0.70)
  Week 8: number analyzed (Participants) | 106 | 100
  Week 8 | 0.1 (0.36) | 0.2 (0.47)
  Week 12: number analyzed (Participants) | 102 | 94
  Week 12 | 0.1 (0.38) | 0.1 (0.38)
  Endpoint | 0.3 (0.75) | 0.3 (0.73)

25. Secondary Outcome: Current Opioid Misuse Measures (COMM) Total Scores During Both the Open-Label Titration and Double-Blind Treatment Periods
Description: The COMM was a clinician rated scale developed as a brief self report measure of current aberrant drug-related behavior for patients with chronic pain who were already on long term opioid therapy. A total score was calculated as the sum of the 17 questions. The total score ranged from 0 to 68. A score of 0 indicates no aberrant drug-related behaviors were seen. Patients with a total score of 9 or greater were classified as exhibiting aberrant drug-related behavior.
  The COMM was to be performed at visits 2 and 7 (beginning and end of Open-label Titration period) and weeks 1, 4, 8, and 12 (Double-blind Treatment period) or early termination.
Time Frame: as for outcome 24
Population: Full analysis set. Participants contributing to each time point are included in the number analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo (Double-blind Treatment Period) | Hydrocodone ER (Double-blind Treatment Period)
Number analyzed (Participants) | 147 | 146
units on a scale
  Baseline Open-Label Titration: number analyzed (Participants) | 146 | 146
  Baseline Open-Label Titration | 3.7 (4.10) | 4.2 (4.14)
  Baseline Double-blind Treatment | 3.7 (4.12) | 3.9 (4.29)
  Week 1: number analyzed (Participants) | 136 | 131
  Week 1 | 2.9 (3.70) | 3.1 (3.10)
  Week 4: number analyzed (Participants) | 115 | 111
  Week 4 | 2.4 (3.10) | 2.8 (3.31)
  Week 8: number analyzed (Participants) | 106 | 100
  Week 8 | 2.5 (3.51) | 2.2 (2.87)
  Week 12: number analyzed (Participants) | 102 | 93
  Week 12 | 2.8 (3.51) | 3.0 (3.53)
  Endpoint | 3.0 (3.67) | 3.3 (3.78)

26. Secondary Outcome: Change From Baseline to Endpoint in the Double-Blind Treatment Phase in Electrocardiogram (ECG) Parameters
Description: A 12-lead ECG was conducted at baseline and the last visit during the double-blind treatment period (week 12, or early termination).
Time Frame: Baseline (end of Open-Label Titration Period), Endpoint (last visit up to Week 12) of the Double-blind treatment period
Population: FAS of participants contributing baseline and endpoint data.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Placebo (Double-blind Treatment Period) | Hydrocodone ER (Double-blind Treatment Period)
Number analyzed (Participants) | 146 | 142
msec
  PR interval | -1.8 (16.27) | -2.4 (29.30)
  QRS interval | -0.1 (15.96) | 0.6 (10.43)
  QT interval | -3.1 (27.08) | 2.2 (28.28)
  QTc interval (Bazett) | -1.0 (20.34) | 4.2 (22.74)
  QTc interval (Fridericia) | -2.5 (21.10) | 2.9 (21.70)

ADVERSE EVENTS:
Time Frame: Day 1 up to Day 52 in Open-Label Titration; Day 1 up to Day 128 in Double-Blind Treatment period
Arm/Group | Hydrocodone ER (Open-Label Titration Period) | Placebo (Double-blind Treatment Period) | Hydrocodone ER (Double-blind Treatment Period)
Serious Adverse Events (participants affected / at risk) | 2/389 | 3/147 | 3/146
Other Adverse Events (participants affected / at risk) | 167/389 | 24/147 | 45/146
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydrocodone ER (Open-Label Titration Period) (N=389) | Placebo (Double-blind Treatment Period) (N=147) | Hydrocodone ER (Double-blind Treatment Period) (N=146)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Hernia obstructive (General disorders) | 0 (0) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2) | 0 (0)
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydrocodone ER (Open-Label Titration Period) (N=389) | Placebo (Double-blind Treatment Period) (N=147) | Hydrocodone ER (Double-blind Treatment Period) (N=146)
Constipation (Gastrointestinal disorders) | 55 (61) | 7 (8) | 19 (19)
Nausea (Gastrointestinal disorders) | 70 (75) | 9 (11) | 19 (20)
Vomiting (Gastrointestinal disorders) | 25 (26) | 5 (6) | 9 (9)
Dizziness (Nervous system disorders) | 22 (23) | 1 (1) | 3 (3)
Headache (Nervous system disorders) | 43 (50) | 8 (8) | 10 (13)
Somnolence (Nervous system disorders) | 45 (51) | 1 (1) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 20 (23) | 1 (1) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.